CLINICAL TRIAL: NCT01499238
Title: Comparison of Nasal CPAP and Nasal SIMV in Transient Tachypnea of Newborn
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Principal Investigator, Gamze Demirel, Zekai Tahir Burak Maternity Teaching Hospital, Zekai Tahir Burak Women's Health Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4
Record Dates: First submitted 2011-12-14; First posted 2011-12-26 (Estimated); Last update posted 2011-12-26 (Estimated); Status verified 2011-12

CONDITIONS: Transient Tachypnea of Newborn
Keywords: Efficacy; safety; nasal SIMV; nasal CPAP; infants who are >35 gestational week with wet lung
MeSH Terms: conditions — Transient Tachypnea of the Newborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nasal SIMV (Active Comparator): rate: 30-50/min, PIP: 16, PEEP: 4-6, fİO2: 40%
  Interventions: Device: Nasal SIMV
- nasal CPAP (Active Comparator): PEEP: 4-6 mmHg, Fio2: 40%
  Interventions: Device: nasal CPAP

INTERVENTIONS:
Device: Nasal SIMV — rate: 30-50/min, PIP: 16-20, PEEP: 4-6, FİO2: 40%
  Other Names: nasal SIMV, SLE 5000
  Arms: nasal SIMV
Device: nasal CPAP — PEEP: 4-6 mmHg, FİO2: 40%
  Other Names: NASAL CPAP, SLE 5000
  Arms: nasal CPAP

SUMMARY:
The investigators aimed to compare the efficacy of nasal SIMV and nasal CPAP in patients with wet lung.

DETAILED DESCRIPTION:
We aimed to compare two types of ventilatory support in cases of transient tachypnea of newborn who are >35 gestational week.

ELIGIBILITY:
Inclusion Criteria:

* >35 gestational week
* wetlung

Exclusion Criteria:

* major congenital anomalies

Ages: 2 Hours to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-02 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
efficacy of nasal SIMV and nasal CPAP in infants with wet lung who are >35 weeks gestational age | 3 months

SECONDARY OUTCOMES:
Complications of respiratory support, respiratory insufficiency | 3 months
  pneumothorax

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Demirel, MD, Principal Investigator — Zekai Tahir Burak Women's Health Research and Education Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Zekai Tahir Burak Maternity Teaching Hospital, Ankara, Ankara
  - Zekai Tahir Burak Maternity Teaching Hospital, Division of Neonatology, Ankara